CLINICAL TRIAL: NCT06878976
Title: An Open-Label Study to Assess the Long-term Safety and Efficacy of Solriamfetol in Adults With Binge Eating Disorder
Brief Title: Open-Label Safety Study of Solriamfetol in Subjects With Binge Eating Disorder
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Axsome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOL-BED-303
Record Dates: First submitted 2025-03-14; First posted 2025-03-17 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Binge-Eating Disorder
Keywords: Binge eating disorder; BED; Solriamfetol; Sunosi; Axsome; Non-stimulant therapy; Dopamine norepinephrine reuptake inhibitor; Trace amine-associated receptor 1 (TAAR1) agonist
MeSH Terms: conditions — Binge-Eating Disorder | interventions — solriamfetol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Solriamfetol (Experimental): Up to 52 weeks.
  Interventions: Drug: Solriamfetol 75mg, 150 mg, or 300 mg

INTERVENTIONS:
Drug: Solriamfetol 75mg, 150 mg, or 300 mg — Taken once daily.

SUMMARY:
This is a Phase 3, multi-center, open-label study to evaluate the long-term safety and efficacy of solriamfetol in the treatment of binge eating disorder (BED) in adults.

DETAILED DESCRIPTION:
Eligible subjects will have previously completed the SOL-BED-301 (ENGAGE) study.

This study consists of a Baseline Visit, a 2-week Titration Phase, and a 50-week Maintenance Phase, followed by a 1-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Completion of the treatment period in Study SOL-BED-301.
* Able to comply with study procedures.

Exclusion Criteria:

* Significant change in vital signs, medical history or concomitant medications since enrolling in the SOL-BED-301 study which, in the opinion of the Investigator or the Medical Monitor, would render the subject unsuitable to receive solriamfetol or participate in the study.

Ages: 18 Years to 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Long-term Safety | Up to 52 weeks.
  Incidence of treatment-emergent adverse events following dosing with solriamfetol

CONTACTS AND LOCATIONS:
Locations (29):
- United States (29):
  - Clinical Research Site, Encino, California
  - Clinical Research Site, Long Beach, California
  - Clinical Research Site, Santa Ana, California
  - Clinical Research Site, Walnut Creek, California
  - Clinical Research Site, West Covina, California
  - Clinical Research Site, Cromwell, Connecticut
  - Clinical Research Site, Fort Myers, Florida
  - Clinical Research Site, Hialeah, Florida
  - Clinical Research Site, Jacksonville, Florida
  - Clinical Research Site, Lauderhill, Florida
  - Clinical Research Site, Miami, Florida
  - Clinical Research Site, Orlando, Florida
  - Clinical Research Site, Marietta, Georgia
  - Clinical Research Site, Overland Park, Kansas
  - Clinical Research Site, Boston, Massachusetts
  - Clinical Research Site, Saint Charles, Missouri
  - Clinical Research Site, Cherry Hill, New Jersey
  - Clinical Research Site, Mount Kisco, New York
  - Clinical Research Site, New York, New York
  - Clinical Research Site, Raleigh, North Carolina
  - Clinical Research Site, Cincinnati, Ohio
  - Clinical Research Site, Mason, Ohio
  - Clinical Research Site, North Canton, Ohio
  - Clinical Research Site, Portland, Oregon
  - Clinical Research Site, North Charleston, South Carolina
  - Clinical Research Site, Memphis, Tennessee
  - Clinical Research Site, Austin, Texas
  - Clinical Research Site, Dallas, Texas
  - Clinical Research Site, San Antonio, Texas

REFERENCES:
- See also: Axsome Therapeutics Website — http://www.axsome.com